CLINICAL TRIAL: NCT06072313
Title: Efficacy of Monopolar Dielectric Diathermy and Therapeutic Exercise on Pain, Functionality, Movement Phobia and Quality of Life in Patients With Chronic Neck Pain.
Brief Title: Monopolar Dielectric Diathermy and Therapeutic Exercise on Chronic Neck Pain and Therapeutic Exercise on Pain, Functionality, Movement Phobia on Pain, Functionality, Movement Phobia and Quality of Life of Patients of Patients With Chronic Neck Pain. Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Ph.D., Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UALBIO2022/019
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Neck Pain
Keywords: monopolar electrical diathermy; therapeutic exercise
MeSH Terms: conditions — Chronic Pain; Neck Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monopolar electrical diathermy plus therapeutic yoga (Experimental): The Experimental Group formed by 30 subjects will receive two sessions per week of monopolar electrical diathermy by radiofrequency emission (MDR) by means of the Physicalm® device (device developed by Biotronic Advance Develops SL), and one session of therapeutic neck yoga per week. Diathermy is applied by means of rotational and translational movements, adapting to the muscular fibers of the cervical area, with a pulsed emission of 840 KHz AND 30v dynamically during a treatment time of 20 minutes.
  Interventions: Other: Therapeutic Exercise
- Therapeutic Exercise (Active Comparator): The Control Group formed by 30 subjects will be administered a supervised therapeutic exercise with the same protocol of postures and sequences as in the Experimental Group, but for three days a week. The duration of the sessions will be 60 minutes.
  The yoga program will be designed specifically for people who have chronic neck pain and no previous experience with therapeutic exercise. Classes will be led by a certified Iyengar yoga instructor and physical therapist. The exercise program will consist of standing, seated and supine postures, starting with simple postures and moving on to more complex ones. Props such as belts, blocks, and blankets will be used to enhance safety and alignment. Participants will be asked to focus on their posture, joint positions, and muscle tension in each exercise posture. No formal breathing techniques will be used, but participants will be instructed to align their breath with their movements.
  Interventions: Other: Monopolar electrical diathermy plus therapeutic exercise

INTERVENTIONS:
Other: Monopolar electrical diathermy plus therapeutic exercise — The Experimental Group will undergo two sessions per week of monopolar electrical diathermy by radiofrequency emission (MDR) using the Physicalm® device and one session of therapeutic neck exercise per week.
  Arms: Therapeutic Exercise
Other: Therapeutic Exercise — The exercise program will consist of standing, seated and supine postures, starting with simple postures and moving on to more complex ones. Participants will be asked to focus on their posture, joint positions and muscle tension in each exercise posture.
  Arms: Monopolar electrical diathermy plus therapeutic yoga

SUMMARY:
The aim of this study is to compare the effects of applying monopolar dielectric radiofrequency diathermy plus therapeutic neck yoga with performing only therapeutic neck yoga in patients with non-specific chronic neck pain.

DETAILED DESCRIPTION:
Chronic non-specific neck pain (CNNP) is a widespread public health problem in the modern world. CNNP is considered persistent neck pain or severe neck discomfort for more than 3 months, which is caused by poor posture and mechanical and degenerative changes, excluding pain due to neck cancer, infections, hernias or other neck disorders or pathologies. In the general population, 71% of adults have neck pain at some time in their lives, and its annual prevalence in the general and working population varies between 30% and 50%. In addition, CNNP is an important cause of work absenteeism and disability.

The research of effective techniques and therapies in the approach of this ailment is a current need within the field of physiotherapy and would mean a reduction of the direct and indirect costs in the health systems generated by patients diagnosed with non-specific chronic neck pain. One of the therapies that is achieving positive results in the symptomatology of different musculoskeletal pathologies such as fibromyalgia syndrome , multiple sclerosis or femoropatellar pain syndrome, is the technique of applying monopolar electric diathermy by radiofrequency emission (MDR), using the Physicalm® device which produces an increase in local temperature due to the action of electromagnetic waves that stimulate tissue metabolism and reduce pain.

Due to all the structural and functional alterations that occur in CNNP, within clinical practice guidelines exercise is one of the most important components in rehabilitation programs for patients with neck pain. Recently, supervised therapeutic exercise has been included as a common intervention in clinical practice worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 30 and 65 years of age.
* Diagnosed by a specialist physician of chronic cervical pain of non-specific origin.
* Acceptance and signature of informed consent for voluntary participation in the research study.
* Not to be undergoing any type of physical therapy or pharmacological treatment.
* Acceptance to attend the treatment sessions of the present research study.

Exclusion Criteria:

* Being under rehabilitation or pharmacological treatment of lumbar pathology.
* Alterations of sensitivity or coagulation.
* Thermal sensitivity problems.
* Present osteosynthesis material at lumbar level.
* Present cardiac, epilepsy or tumor complications.
* Non-acceptance of the informed consent or non-attendance to all the sessions that make up the treatment.

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Neck disability index | Change from baseline disability at four weeks and three months
  The neck disability index consists of 10 questions addressing functional activities such as personal care, lifting, reading, work, driving, sleeping, recreational, pain intensity, concentration and headache.
Active and Latent Myofascial Trigger Points (Number of trigger Points) | Change from baseline myofascial trigger points at four weeks and three months
  Myofascial Trigger Points will be explored in the following pairs of muscles: occipital, splenius capitis, sternocleidomastoid, scalene, trapezius, supraspinatus, infraspinatus, and multifidus.

SECONDARY OUTCOMES:
Pain (Visual Analog Scale) | Change from baseline pain intensity at four weeks and three months
  Pain will be assessed with the Visual Analog Scale (VAS), which assesses the pain intensity and degree of relief experienced by the patient (scored of 0 = no pain; 10 = unbearable pain).
McGill Pain Questionnaire | Change from baseline pain intensity at four weeks and three months
Quality of Life (SF-36 quality of life questionnaire) | Change from baseline quality of life at four weeks and three months
  The SF-36 quality of life questionnaire assesses 8 domains including physical functioning, physical role, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.
Quality of Sleep (Pittsburgh Quality of Sleep Questionnaire Index) | Change from baseline quality of sleep at four weeks and three months
  The Pittsburgh Quality of Sleep Questionnaire Index (PSQI) will be used to study the quality of sleep. It comprises 24 items where the subjects respond to 19 of these items, and individual living in the same dwelling (or hospital room) responds to the remaining 5. Scores are obtained on each of 7 components of sleep quality: subjective quality, sleep latency, sleep duration, habitual sleep efficacy, sleep perturbations, use of hypnotic medication, and daily dysfunction.
Cervical Range of Motion | Change from baseline range of motion at four weeks and three months
  Cervical range of motion is assessed with the patient sitting comfortably on a chair, with both feet flat on the floor, hips and knees at 90º of flexion, and buttocks positioned against the back of the chair.
Tampa scale for kinesiophobia | Change from baseline phobia of movement at four weeks and three months
  The 17-item Tampa scale for kinesiophobia assesses fear of movement or of injury or reinjury.

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaida María Castro Sánchez, Almería, Almeria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vassilaki M, Hurwitz EL. Insights in public health: perspectives on pain in the low back and neck: global burden, epidemiology, and management. Hawaii J Med Public Health. 2014 Apr;73(4):122-6. No abstract available. PMID 24765562
- [Background] Hogg-Johnson S, van der Velde G, Carroll LJ, Holm LW, Cassidy JD, Guzman J, Cote P, Haldeman S, Ammendolia C, Carragee E, Hurwitz E, Nordin M, Peloso P. The burden and determinants of neck pain in the general population: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S46-60. doi: 10.1016/j.jmpt.2008.11.010. PMID 19251074
- [Background] Monticone M, Iovine R, de Sena G, Rovere G, Uliano D, Arioli G, Bonaiuti D, Brugnoni G, Ceravolo G, Cerri C, Dalla Toffola E, Fiore P, Foti C; Italian Society of Physical and Rehabilitation Medicine (SIMFER). The Italian Society of Physical and Rehabilitation Medicine (SIMFER) recommendations for neck pain. G Ital Med Lav Ergon. 2013 Jan-Mar;35(1):36-50. PMID 23798233
- [Background] Strine TW, Hootman JM. US national prevalence and correlates of low back and neck pain among adults. Arthritis Rheum. 2007 May 15;57(4):656-65. doi: 10.1002/art.22684. PMID 17471542
- [Background] US Burden of Disease Collaborators; Mokdad AH, Ballestros K, Echko M, Glenn S, Olsen HE, Mullany E, Lee A, Khan AR, Ahmadi A, Ferrari AJ, Kasaeian A, Werdecker A, Carter A, Zipkin B, Sartorius B, Serdar B, Sykes BL, Troeger C, Fitzmaurice C, Rehm CD, Santomauro D, Kim D, Colombara D, Schwebel DC, Tsoi D, Kolte D, Nsoesie E, Nichols E, Oren E, Charlson FJ, Patton GC, Roth GA, Hosgood HD, Whiteford HA, Kyu H, Erskine HE, Huang H, Martopullo I, Singh JA, Nachega JB, Sanabria JR, Abbas K, Ong K, Tabb K, Krohn KJ, Cornaby L, Degenhardt L, Moses M, Farvid M, Griswold M, Criqui M, Bell M, Nguyen M, Wallin M, Mirarefin M, Qorbani M, Younis M, Fullman N, Liu P, Briant P, Gona P, Havmoller R, Leung R, Kimokoti R, Bazargan-Hejazi S, Hay SI, Yadgir S, Biryukov S, Vollset SE, Alam T, Frank T, Farid T, Miller T, Vos T, Barnighausen T, Gebrehiwot TT, Yano Y, Al-Aly Z, Mehari A, Handal A, Kandel A, Anderson B, Biroscak B, Mozaffarian D, Dorsey ER, Ding EL, Park EK, Wagner G, Hu G, Chen H, Sunshine JE, Khubchandani J, Leasher J, Leung J, Salomon J, Unutzer J, Cahill L, Cooper L, Horino M, Brauer M, Breitborde N, Hotez P, Topor-Madry R, Soneji S, Stranges S, James S, Amrock S, Jayaraman S, Patel T, Akinyemiju T, Skirbekk V, Kinfu Y, Bhutta Z, Jonas JB, Murray CJL. The State of US Health, 1990-2016: Burden of Diseases, Injuries, and Risk Factors Among US States. JAMA. 2018 Apr 10;319(14):1444-1472. doi: 10.1001/jama.2018.0158. PMID 29634829
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Cote P, van der Velde G, Cassidy JD, Carroll LJ, Hogg-Johnson S, Holm LW, Carragee EJ, Haldeman S, Nordin M, Hurwitz EL, Guzman J, Peloso PM. The burden and determinants of neck pain in workers: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S70-86. doi: 10.1016/j.jmpt.2008.11.012. PMID 19251078
- [Background] Kjellman G, Skargren E, Oberg B. Prognostic factors for perceived pain and function at one-year follow-up in primary care patients with neck pain. Disabil Rehabil. 2002 May 10;24(7):364-70. doi: 10.1080/10.1080/09638280110101532. PMID 12022786
- [Background] Hurwitz EL, Carragee EJ, van der Velde G, Carroll LJ, Nordin M, Guzman J, Peloso PM, Holm LW, Cote P, Hogg-Johnson S, Cassidy JD, Haldeman S; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Treatment of neck pain: noninvasive interventions: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S123-52. doi: 10.1097/BRS.0b013e3181644b1d. PMID 18204386
- [Background] Ibanez-Vera AJ, Garcia-Romero JC, Alvero-Cruz JR, Lomas-Vega R. Effects of Monopolar Dielectric Radiofrequency Signals on the Symptoms of Fibromyalgia: A Single-Blind Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Apr 3;17(7):2465. doi: 10.3390/ijerph17072465. PMID 32260313
- [Background] Hochsprung A, Escudero-Uribe S, Ibanez-Vera AJ, Izquierdo-Ayuso G. Effectiveness of monopolar dielectric transmission of pulsed electromagnetic fields for multiple sclerosis-related pain: a pilot study. Neurologia (Engl Ed). 2021 Jul-Aug;36(6):433-439. doi: 10.1016/j.nrleng.2018.03.003. Epub 2020 Feb 7. PMID 34238526
- [Background] Albornoz-Cabello M, Ibanez-Vera AJ, Aguilar-Ferrandiz ME, Espejo-Antunez L. Monopolar dielectric diathermy by emission of radiofrequency in Patellofemoral pain. A single-blind-randomized clinical trial. Electromagn Biol Med. 2020 Oct 1;39(4):282-289. doi: 10.1080/15368378.2020.1793169. Epub 2020 Jul 19. PMID 32683992
- [Background] Albornoz-Cabello M, Ibanez-Vera AJ, De la Cruz-Torres B. Efficacy of monopolar dielectric transmission radio frequency in panniculus adiposus and cellulite reduction. J Cosmet Laser Ther. 2017 Nov;19(7):422-426. doi: 10.1080/14764172.2017.1342041. Epub 2017 Jul 5. PMID 28678582
- [Background] Kumaran B, Watson T. Skin thermophysiological effects of 448 kHz capacitive resistive monopolar radiofrequency in healthy adults: A randomised crossover study and comparison with pulsed shortwave therapy. Electromagn Biol Med. 2018;37(1):1-12. doi: 10.1080/15368378.2017.1422260. Epub 2018 Jan 8. PMID 29308927
- [Background] 17. Kumaran, B., Herbland, A., Watson, T. 2017. Continuous mode 448 kHz capacitive resistive monopolar radiofrequency induces greater deep blood flow changes compared to pulsed mode shortwave: A crossover study in healthy adults. Eur. J. Physiotherapy 19:137-46.
- [Background] Kay TM, Gross A, Goldsmith C, Santaguida PL, Hoving J, Bronfort G; Cervical Overview Group. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD004250. doi: 10.1002/14651858.CD004250.pub3. PMID 16034925
- [Background] Gross AR, Paquin JP, Dupont G, Blanchette S, Lalonde P, Cristie T, Graham N, Kay TM, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Santaguida PL, Yee AJ, Radisic GG, Hoving JL, Bronfort G; Cervical Overview Group. Exercises for mechanical neck disorders: A Cochrane review update. Man Ther. 2016 Aug;24:25-45. doi: 10.1016/j.math.2016.04.005. Epub 2016 Apr 20. PMID 27317503
- [Background] Feuerstein G. The Yoga Tradition. Prescott, AZ, USA: Hohm Press, 1998.
- [Background] Cramer H, Lauche R, Langhorst J, Dobos G. Is one yoga style better than another? A systematic review of associations of yoga style and conclusions in randomized yoga trials. Complement Ther Med. 2016 Apr;25:178-87. doi: 10.1016/j.ctim.2016.02.015. Epub 2016 Mar 3. PMID 27062966
- [Background] Bramberg EB, Bergstrom G, Jensen I, Hagberg J, Kwak L. Effects of yoga, strength training and advice on back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2017 Mar 29;18(1):132. doi: 10.1186/s12891-017-1497-1. PMID 28356091
- [Background] Rajalaxmi V, Jasim A, Sudhakar S, et al. To analyse the effectiveness of yoga, pilates and Tai Chi exercise for chronic mechanical neck pain-a randomized controlled trail. Biomedicine 2018;38:156-60.